CLINICAL TRIAL: NCT04262778
Title: Diagnostic Accuracy of Electrochemical Skin Conductance Measurement in Paediatric Small Fibre Neuropathy Following Neurotoxic Chemotherapy
Brief Title: Diagnostic of Chemotherapy Induced Neuropathy in Children
Acronym: SUDOPED
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Société Française de lutte contre les cancers et leucémies de l'enfant et de l'adolescent (SFCE) (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190700; 2019-A03044-53 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-01-31; First posted 2020-02-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Chemotherapy induced peripheral neuropathy (CIPN); child; outcome; electrochemical skin conductances (ESC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: electrochemical skin conductance measurement — electrochemical skin conductance measurement

SUMMARY:
The purpose of this study is to determine the diagnostic accuracy of a newly developed tool (Electrochemical Skin Conductances (ESC) measurement) easy-to-perform, non-invasive, highly reproductible and not requiring specific training, to identify pediatric chemotherapy-induced-peripheral-neuropathies (CIPN). CIPN are a frequent (20 to 75% depending on the drug), early and potentially severe long-lasting and dose limiting adverse effect of treatments in immuno-hematology and cancerology. The pathophysiology, the chronology of injury (ie small then large sensory nerve fiber or vice-versa) and the age-related short/long-term impact on peripheral nerves remain largely not understood. Clinical signs of CIPN are highly heterogenous, often under-recognized and include diverse sensory symptoms and pain. Persistent loss of sensation and strength as well as neuropathic pain may have a short/long-term impact in term of functional limitations and quality of life. There is a lack of specific and sensitive measurement tools for CIPN in the pediatric population. Neurophysiological tools (except electro-neuro-myography allowing only the assessment of large myelinated nerves) are not implemented in the pediatric oncology-hematology everyday practice: they are often invasive and/or poorly reproducible, not accessible for "bedside" follow-up, and lacking normative values, thus often dedicated only to research. ESC may provide an early and quantitative assessment of small fiber dysfunction in children, a prerequisite for the identification of additional preventive or curative approaches in CIPN.

DETAILED DESCRIPTION:
Epidemiology and suggested mechanisms involved in pediatric chemotherapy induced neuropathy: Pediatric chemotherapy induced peripheral neuropathy (CIPN) is an early (often occurring within the first three months), potentially severe long-lasting and dose limiting adverse effect of treatment in immuno-hematology and cancerology. It constitutes the second most common cause of dose limitation compromising therapy efficacy after hematological adverse effects. Expanding number of potentially toxic treatment for the peripheral nervous system are currently used. Peripheral nerve toxicity has been mainly described with the platinum-based antineoplastics (particularly oxaliplatin and cisplatin), vinca-alkaloids (particularly vincristine and vinblastine), taxanes (paclitaxel, docetaxel), proteasome inhibitors (bortezomib) and immunomodulatory drugs (thalidomide). Vinca-alkaloids are used for treatment of acute leukemia, lymphoma, various solid tumors and are responsible for neuropathy of any grade (National Cancer Institute Common Terminology Criteria for Adverse Effects, NCI-CTAE grade 1 to 4) in 75-100% of patients, including 10-52% grade 3/4 neuropathy with probable dose-toxicity relationship. Platinum compounds (Cisplatin, Carboplatin, Oxaliplatin) are used for the treatment of various solid tumors. Cisplatin and Carboplatin are often used in combination therapy with Vincristine making it difficult to appreciate its relative contribution to peripheral toxicity. Oxaliplatin peripheral neurotoxicity is observed in 37-50% and 3-8% of patients for Common Terminology Criteria for Adverse Effects (CTAE) grade 1/2 and grade 3/4 respectively. Bortezomib is used for preventing antibody mediated in transplantation and for others autoimmune diseases. Thalidomide is used for the treatment of diverse inflammatory conditions such as refractory inflammatory bowel disease, juvenile rheumatoid arthritis and vasculitis and is associated with peripheral neuropathy in 20-40% (Grade > = 2). Clinical features of CIPN are heterogeneous but sensory nerves involvement is prominent. In a very recent study, 23,5% of patients presented with a decrease in sural sensory nerve amplitude several years after exposure of neurotoxic chemotherapy, suggesting a long-term impact with an irreversible reduction of functioning axons. Various molecular and cellular mechanisms have been suggested. Indeed, chemotherapy treatments result in changes to cellular structure and function including alteration in voltage gate ion channels, neurotransmission, organelle function and intracellular signalling. For example, putative mechanisms involved in the development of vincristine-induced peripheral neuropathy are highly multifactorial and depending on disease and patient factors (age, genetic alterations in pharmacokinetic/pharmacodynamic pathways, and susceptibility to hereditary neuropathy). Possible effects of vincristine on tubulin polymerization leading to microtubule destabilization and deficit in axonal transport may be the main mechanisms contributing to the development of vincristine-induced CIPN. Although the individual biological eﬀects of these drugs on cancer cells are relatively well known and studied extensively, the age-related short- and long-term impact on peripheral nerves, prerequisite for the identification of additional preventive or curative approaches, remains incompletely understood.

-Diagnosis and management of pediatric chemotherapy induced neuropathy: Symptoms of neurotoxicity induced by chemotherapy in the peripheral nerve system are often under-recognized and undiagnosed. One major reason has been the lack of specific and sensitive measurement tools for CIPN in the pediatric population. Clinical signs of CIPN are highly heterogenous and include sensory symptoms, including paresthesia (tingling, numbness), dysesthesia, allodynia, hyperalgesia, hypoalgesia or pain (burning/shooting sensation, electric-shock-like). Clinical manifestations could be related to dysfunction of small sensory nerve fibers causing allodynia or hyperpathia. The younger the patient, the less specific the complaints may be. Patients may manifest behavior troubles or refuse to move or to be touched (4). Furthermore, little is known about the long-term impact of CIPN in survivors of childhood cancer in term of quality of life, sleep disorders, psychopathological disorders and learning skills. There is also currently no evidence-based preventive and treatment strategy for CIPN in children. Drugs used in routine clinical practice are those that are efficient in other neuropathic conditions including tricyclic antidepressant, GABAergic agents. However, systemic adverse effects of these treatments are frequent, and the control of the neuropathic pain remains to be optimized. The most commonly used assessment scale for CIPN is the CTCAE, rating 0 to 5 the severity of the sensory or motor neuropathy. CTCAE, although easy to use, displays a poor interobserver agreement and do not provide the specific clinical characteristics of CIPN. In recent years, the Total Neuropathy Scale (TNS) was developed as clinical assessment of peripheral neuropathy in adults and has demonstrated reliability and validity in measuring CIPN in adult cancer patient. The pediatric modified Total Neuropathy Scale (Ped-mTNS) has been developed and tested in population of children (for patient age above 5 years) with cancer with acceptable interrater reliability, test retest reliability and internal consistency. The Ped-mTNS has 5 clinical testing domains: light touch sensation, pin sensibility, vibration sensibility, strength, and deep tendon reflexes. The most widely agreed method for diagnosing small fiber neuropathy is skin biopsy. Intraepidermal nerve ﬁber density (IENFD) assessment via skin biopsies, which evaluates the epidermal loss of Aδ/C small ﬁber, cannot be used for follow-up in current practice due to its invasiveness, delay in obtaining results. Furthermore, normal values are lacking in children. Various neurophysiological methods are available in adult for detecting CIPN. Nerve conduction studies (NCS) allows only the assessment of large myelinated nerves and therefore are not suitable for non-myelinated small ﬁber assessment. In addition, specialized tool are used for the exploration of small non-myelinated fibers including, quantified exploration of the thermal sensitivity (Quantitative Sensory Testing assessing sensory C fibers), laser evoked potentials (PEL assessing sensory A-delta fibers), quantitative Sudomotor Axon Reﬂex Testing (QSART) assessing small ﬁber impairment via sudomotor function.

All these tools are not implemented in the pediatric current clinical practice because they are either reserved for research, or technically challenging to perform. or invasive, or poorly reproducible, or lacking normal values. These methods are not accessible to pediatric oncologists and not suitable for follow up patients during chemotherapy.

-Longitudinal assessment of CIPN by the measurement of electrochemical skin conductances (ESC) by SUDOSCAN® (Impeto Medical, Paris, France) Among the small fibers, those innervating the sweat glands degenerate after toxic injury, and are the first to regenerate if the toxic injury is removed. Thus, the fibers innervating the sweat glands could be considered a good marker of small fibers injuries. A new device has been recently developed to quantify the sudomotor function, quickly, non-invasively and quantitatively. The technique is based on the measurement of an electrical signal produced by an electrochemical reaction between the chloride ions present in the sweat and stainless-steel electrodes at which a low current (< 4 V) is applied. The device automatically calculates ESC, expressed in microSiemens (µS), as the ratio between the current generated and the constant direct current stimulus applied to the electrodes. ESC is thought to reflect the innervation of cutaneous sweat glands (autonomic unmyelinated nerve fibres) containing functional chloride channels. In adult, several studies have validated the method and evaluated its diagnostic accuracy to detect small fiber dysfunction in diverse conditions, including diabetes, Familial Transthyretin Amyloid Polyneuropathy, Fabry disease, toxic neuropathy…etc. This method has been compared to reference methods assessing small fiber dysfunction and its diagnostic performance has been evaluated in comparison with the gold standard IENFD. Furthermore, the diagnostic sensitivity for detecting small-fiber neuropathies of ESC measurements was compared to four other neurophysiological tests in 87 adult patients with clinically defined (n = 33) or possible (n = 54) small-fiber neuropathy. The neurophysiological tests, performed at the four extremities (hands and feet), included a quantified study of the thermal sensitivity, with determination of the detection of warm and cold thresholds (WDT and CDT), the recording of evoked potentials by laser stimulation (ELP) and Sympathetic Skin Responses (SSR) and measurement of ESCs. ELPs were the most sensitive test (modified in 56/71 patients with at least one abnormal test (79%)), followed by ESCs (61%), WDT (55%), SSR (41%) and finally the CDT (29%). Thus, in adult, the combination of PEL, assessing sensory A-delta fibers of WDT assessing sensory C fibers, and ESCs, evaluating autonomous C fibers, seems to represent a relevant approach for the diagnosis of SFN. The ELP, although technically efficient, still has some disadvantages, such as the cost of the equipment, the duration of the examination and the technicity of the recordings, contrarily to ESCs that remains a quick test (3 minutes), easy to do and to interpret and can be used as bedside tool.

To date, no research on using this method in children has been published. Very recently normative values have been established in children. Values observed for ESC measurements in healthy children are similar in all group of age and values observed in healthy adults suggesting that sudomotor nerve maturation occurs very early in life. Thus, ESC measurement may be a quick, reproductible, non-invasive and quantitative assessment of small fiber dysfunction in children.

ELIGIBILITY:
Inclusion Criteria:

* aged 5-17 years
* initiating a potentially neurotoxic chemotherapy alkaloids (vincristine vinblastine, vinorelbine), Platinum compounds (oxaliplatine, cisplatine, carboplatine), proteasome inhibitors (bortezomib), Thalidomide derivatives, taxanes (such as taxol or taxotere), antiCD30 (brentuximab)
* Information of the legal representative of the patient Affiliated to social security regime or an equivalent system

Exclusion Criteria:

* history of peripheric neuropathy
* current antiepileptic medications or other treatment for neurogenic pain (tegretol, neurontin, lyrica, laroxyl, rivotril,… etc)
* distal skin lesions that do not allow electrochemical skin conductance measurement
* child not able to stand during the time of examination

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Child receiving a Potentially Neurotoxic Chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Diagnosis of neuropathy using a ped-mTNS Score | 6 months
  Define as a ped-mTNS score ≥ 5
Diagnosis of neuropathy using electrochemical skin conductance | 6 months
  Define as a mean of electrochemical skin conductance measured at hands and feet < pediatric norms.

SECONDARY OUTCOMES:
Changes in electrochemical skin conductance before clinical signs | 6 months
  Changes in mean of electrochemical skin conductance measured at hands and feet before clinical signs
Changes in electrochemical skin conductance after treatment | 6 months
  Changes in mean of electrochemical skin conductance measured at hands and feet after treatment of neuropathic pain

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Gitiaux, MD PhD, Principal Investigator — Assistance Public Hôpitaux de Paris
Locations (1):
- Necker- enfants maladies hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kandula T, Farrar MA, Kiernan MC, Krishnan AV, Goldstein D, Horvath L, Grimison P, Boyle F, Baron-Hay S, Park SB. Neurophysiological and clinical outcomes in chemotherapy-induced neuropathy in cancer. Clin Neurophysiol. 2017 Jul;128(7):1166-1175. doi: 10.1016/j.clinph.2017.04.009. Epub 2017 Apr 25. PMID 28511129
- [Background] Kandula T, Farrar MA, Cohn RJ, Mizrahi D, Carey K, Johnston K, Kiernan MC, Krishnan AV, Park SB. Chemotherapy-Induced Peripheral Neuropathy in Long-term Survivors of Childhood Cancer: Clinical, Neurophysiological, Functional, and Patient-Reported Outcomes. JAMA Neurol. 2018 Aug 1;75(8):980-988. doi: 10.1001/jamaneurol.2018.0963. PMID 29799906
- [Background] Gilchrist LS, Tanner L. The pediatric-modified total neuropathy score: a reliable and valid measure of chemotherapy-induced peripheral neuropathy in children with non-CNS cancers. Support Care Cancer. 2013 Mar;21(3):847-56. doi: 10.1007/s00520-012-1591-8. Epub 2012 Sep 20. PMID 22993026
- [Background] Gibbons CH, Wang N, Freeman R. Capsaicin induces degeneration of cutaneous autonomic nerve fibers. Ann Neurol. 2010 Dec;68(6):888-98. doi: 10.1002/ana.22126. PMID 21061393
- [Background] Castro J, Miranda B, Castro I, de Carvalho M, Conceicao I. The diagnostic accuracy of Sudoscan in transthyretin familial amyloid polyneuropathy. Clin Neurophysiol. 2016 May;127(5):2222-7. doi: 10.1016/j.clinph.2016.02.013. Epub 2016 Feb 27. PMID 27072093
- [Background] Lefaucheur JP, Wahab A, Plante-Bordeneuve V, Sene D, Menard-Lefaucheur I, Rouie D, Tebbal D, Salhi H, Creange A, Zouari H, Ng Wing Tin S. Diagnosis of small fiber neuropathy: A comparative study of five neurophysiological tests. Neurophysiol Clin. 2015 Dec;45(6):445-55. doi: 10.1016/j.neucli.2015.09.012. Epub 2015 Nov 17. PMID 26596193
- [Background] Leclair-Visonneau L, Bosquet T, Magot A, Fayet G, Gras-Le Guen C, Hamel A, Pereon Y. Electrochemical skin conductance for quantitative assessment of sweat function: Normative values in children. Clin Neurophysiol Pract. 2016 Jul 27;1:43-45. doi: 10.1016/j.cnp.2016.07.001. eCollection 2016. PMID 30214959